CLINICAL TRIAL: NCT02251366
Title: A Multi-Satellite Comparison of Standard-of-Care, Physician-Based Retinal Evaluation Versus Physician-Guided Diagnostic Evaluation in the Management of Neovascular Age-Related Macular Degeneration With Anti-Vascular Endothelial Growth Factor Therapy
Brief Title: NVAMD Satellite Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NA_00088759
Record Dates: First submitted 2014-09-09; First posted 2014-09-29 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Neovascular Age Related Macular Degeneration
Keywords: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SOC Examination Based Cohort (No Intervention): Participants in this arm will receive standard of care (SOC) retinal examinations at each study visit.
- Physician-Guided Diagnostic (Active Comparator): Participants in this arm of the study will only receive the physical standard-of-care retinal examination at the 4-month and -month office visits, unless requested by the Physician-Investigator or study participant. At each standard study visit, the physician will use diagnostic imaging to determine if the participant will receive the anti-VEGF injection.
  Interventions: Procedure: Physician-guided diagnostic

INTERVENTIONS:
Procedure: Physician-guided diagnostic — NVAMD participants in the physician-guided diagnostic arm will have receive injections based on diagnostic imaging provided by optical coherence tomography and optional fluorescein angiography, those in this group will only receive retinal examinations at the 4- and 8-month clinic visits.
  Arms: Physician-Guided Diagnostic

SUMMARY:
Intravitreal delivery of anti-vascular endothelial growth factor (VEGF) drugs has revolutionized the management of neovascular age-related macular degeneration (NVAMD). However, the requirement for near monthly administration of therapy coupled with the growing number of patients needing treatment has become a universal challenge in efficient delivery of care for retina physicians. While many retina practices have both increased the size of their staffs to accommodate the growing patient population and increased efficiency with the aid of digital photography, patient encounter times in clinic continue to increase, often spanning 2-4 hours. While maintaining the highest level of patient care, a streamlined alternative in the evaluation of patients with NVAMD to determine whether intravitreal therapy with an anti-VEGF agent is indicated at a particular office visit would be desirable.

This multi-satellite, prospective, randomized pilot study will compare standard-of-care, physician- based retinal evaluation, defined as retinal examination by a physician and standard imaging with optical coherence tomography (OCT) and optional fluorescein angiography (FA), versus physician-guided diagnostic evaluation, defined as standard imaging with OCT and optional FA without retinal examination by a physician in the management of NVAMD with anti-VEGF therapy. Outcomes for this study are aimed primarily at demonstrating that the physician-guided diagnostic approach to managing patients with NVAMD is not inferior to the physician-based retinal evaluation based on measures such as a change from baseline in visual acuity and in central subfield thickness (CSF) on OCT. Other outcomes to be assessed in this study are length of visit times, numbers of intravitreal injections of anti-VEGF agents administered, numbers of diagnostic tests performed to determine whether treatment should be given at each visit, and frequency of retinal examinations performed for each participating patient in each cohort. Perceptions of quality of vision and patient satisfaction will be captured by interviews with patients following each clinic visit; clinical impressions of physicians will be captured by a brief physician survey. Finally, the feasibility of recruiting patients, as measured by how many eligible patients are seen at each Wilmer satellite, how many patients agree to be randomized, how many patients follow-up, and the attrition rates at the 4 and 8-month outcome visits will be assessed.

ELIGIBILITY:
Inclusion criteria:

* Established diagnosis of NVAMD in one or both eyes
* Received 2 or more intravitreal injections of anti-VEGF therapy from the retinal physician during the prior 6 months
* Need for more therapy on a near monthly basis is anticipated
* Usual corrected visual acuity (UCVA) of at least one eye must be 20/200 or better
* Must be physically able to cooperate with OCT and other diagnostic imaging procedures
* Must be able to give informed consent and be able to complete telephone surveys

Exclusion criteria:

* Systemic disease that can affect the peripheral retina (e.g., diabetes mellitus, sickle cell)
* History of symptomatic posterior vitreous detachment, retinal tear, or retinal detachment
* History of retinal surgery will not be enrolled.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
Change in visual acuity from baseline | up to two years
Change in OCT CSF from baseline | up to two years

SECONDARY OUTCOMES:
total encounter time for each arm | up to two years

OTHER OUTCOMES:
Number of intravitreal anti-VEGF injections administered | up to two years
number of diagnostic tests performed | up to two years
number of retinal examinations performed | up to two years

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Solomon, MD, Principal Investigator — Johns Hopkins University
Locations (5):
- United States (5):
  - Wilmer Eye Institute, Bel Air, Maryland
  - Wilmer Eye Institute, Bethesda, Maryland
  - Wilmer Eye Institute, Columbia, Maryland
  - Wilmer Eye Institute, Frederick, Maryland
  - Wilmer Eye Institute, Lutherville, Maryland

REFERENCES:
- [Derived] Solomon SD, Kyerematen V, Qutab M, Wenick AS, Wang J, Hawkins BS. Are Dilated Fundus Examinations Needed for OCT-Guided Retreatment of Exudative Age-Related Macular Degeneration? A Prospective, Randomized, Pilot Study. Clin Ophthalmol. 2021 Aug 12;15:3401-3417. doi: 10.2147/OPTH.S315554. eCollection 2021. PMID 34408396